CLINICAL TRIAL: NCT06102499
Title: Comparison of Pulse Oximetry (SpO2) With Different Oximeters and Arterial Saturation (SaO2): Oxygap2 Study
Acronym: Oxygap 2
Status: Recruiting | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, François Lellouche, Principal Investigator, Laval University
Other Study IDs: 22373
Record Dates: First submitted 2023-10-06; First posted 2023-10-26 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Respiratory Failure; Hypoxemia; Hyperoxemia
MeSH Terms: conditions — Respiratory Insufficiency; Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pediatric population: Pediatric population < 18 years old (estimated 100 patients)
  Interventions: Device: SpO2 and SaO2 comparison
- Adult population: Adult population >or= 18 years old (estimated 100 patients)
  Interventions: Device: SpO2 and SaO2 comparison

INTERVENTIONS:
Device: SpO2 and SaO2 comparison — Several pulse oximeter will be place on patient find few minutes before arterial blood gases. During an arterial blood sample, all SpO2 will be recorded

SUMMARY:
The oximeter is used to monitor intensive care patients undergoing oxygen therapy. It indicates pulsed oxygen saturation (SpO2), a reflection of arterial oxygen saturation (SaO2) which enables detection of hypoxemia and hyperoxia, both deleterious state. Current SpO2 recommendations aim to reduce both risk of hypoxemia and hyperoxia. SpO2 is considered the 5th vital sign.

Current recommendations for SpO2 targets do not consider the variability of oximeters used in clinical practice. This variability and lack of specification represent an obstacle to an optimal practice of oxygen therapy.

Thus, this study aims to compare the SpO2 values of different oximeters (General Electric-GE, Medtronic, Masimo and Nonin) used in clinical practice with the SaO2 reference value obtained by an arterial gas in order to specify the precision and the systematic biases of the oximeters studied. This data will also make it possible to refine the recommendations concerning optimal oxygenation

ELIGIBILITY:
Adult population

Inclusion Criteria:

* ≥ 18 years old (adult population) -
* Patients admitted to the Intensive Care Unit
* Artery catheter already installed

Pediatric population

* Below 18 years old
* Patients admitted to the Intensive Care Unit
* Artery catheter already installed

Exclusion Criteria:

* No or poor signal with the usual pulse oximeter/based on clinician judgment
* High dose of vasopressors or inotropes (epinephrine or norepinephrine ˃ 1mcg/kg/min), shock state (lactates above 3 mmoles/L)
* Pigmented nails or nail polish
* Methemoglobinemia history
* Hemoglobin below 80 g/L
* Patient in isolation (multi-resistant bacteria, C-Difficile, SARS-COV-2…)
* Prone position, Extra Corporel Membrane Oxygenator

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patient in ICU with arterial catheter already installed will be consider
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Difference between GE oximeter SpO2 value and the SaO2 value on arterial blood gases | During procedure (arterial blood gas sample collection)
  Difference between GE oximeter SpO2 and the SaO2 value
Difference between Nellcor oximeter SpO2 value and the SaO2 value on arterial blood gases | During procedure (arterial blood gassample collection)
  Difference between Nellcor oximeter SpO2 and the SaO2 value
Difference between Masimo oximeter SpO2 value and the SaO2 value on arterial blood gases | During procedure (arterial blood gas sample collection)
  Difference between Masimo oximeter SpO2 and the SaO2 value
Difference between Nonin oximeter SpO2 value and the SaO2 value on arterial blood gases | During procedure (arterial blood gas sample collection)
  Difference between Nonin oximeter SpO2 and the SaO2 value

SECONDARY OUTCOMES:
Overestimation and underestimation of SaO2 | During procedure (arterial blood gas sample collection)
  Percent of pairs with overestimation and underestimation of SaO2 for each oximeter.
Hypoxemia detection | During procedure (arterial blood gas sample collection)
  Ability to detect hypoxemia (SpO2 below 90% and PaO2 < 60 mmHg)

OTHER OUTCOMES:
Hyperoxemia detection | During procedure (arterial blood gas sample collection)
  Ability to detect hyperoxemia (SpO2 above 95% and PaO2 > 100 mmHg)
Gaps between the different oximeters | During procedure (arterial blood gas sample collection)
  Average of the SpO2 value gaps between the different oximeters tested

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - CHUM, Montreal, Quebec
  - CHU Ste-Justine, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No